CLINICAL TRIAL: NCT00116220
Title: A Phase III Trial of External Beam of Radiotherapy +/- Total Androgen Suppression for High Risk Clinically Organ-Confined Prostate Cancer
Brief Title: Study of External Beam Radiation Therapy With and Without Hormonal Therapy to Treat Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Saint Anne's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Metro West Medical Center (Other)
Responsible Party: Principal Investigator, Anthony V. D'Amico, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95-096
Record Dates: First submitted 2005-06-27; First posted 2005-06-28 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Total Androgen Suppression; endorectal coil MRI; External Beam Radiation Therapy; Prostate Cancer- High Risk, clinically Organ-Confined
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment 1 (Active Comparator): External beam radiation therapy + 6 months total androgen ablation
  Interventions: Drug: Flutamide (Eulexin) and Lupron or Zoladex; Radiation: External Beam Radiotherapy
- Treatment 2 (Active Comparator): External beam radiation therapy
  Interventions: Radiation: External Beam Radiotherapy

INTERVENTIONS:
Drug: Flutamide (Eulexin) and Lupron or Zoladex — Androgen suppression therapy
  Arms: Treatment 1
Radiation: External Beam Radiotherapy — Once a day, 4-5 days per week for approximately 2 months

SUMMARY:
This clinical study was to determine if the use of 6 months of total androgen suppression (hormonal therapy) when added to radiation therapy for localized-high risk prostate cancer would improve overall survival.

DETAILED DESCRIPTION:
This was a randomized study comparing external beam radiation therapy with total androgen ablation for 6 months with radiation therapy alone. Drugs were given 2 months prior, 2 months during, and 2 months after radiation therapy. Eulexin and Lupron or Zoladex was used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate cancer
* Negative bone scan
* Lymph nodes by CT or MRI
* Adequate blood work
* Performance Status - ECOG 0-1
* Life expectancy of at least 10 years
* >40 years of age

Exclusion Criteria:

* Prior history of malignancy
* Prior hormonal therapy or chemotherapy
* Prior pelvic radiation therapy
* Unable to tolerate lying still 5-10 minutes/day

Min Age: 41 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 1995-09; Primary Completion 2001-04 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To determine if the 2 year freedom from PSA failure is increased in patients receiving total androgen suppression and radiation therapy compared to those patients receiving radiation therapy alone. | Years

SECONDARY OUTCOMES:
Evaluate the quality of life of patients receiving total androgen suppression and radiation therapy | Years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony V D'Amico, M.D. Ph.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Background] Taneja SS. Re: Long-Term Follow-up of a Randomized Trial of Radiation with or without Androgen Deprivation Therapy for Localized Prostate Cancer. J Urol. 2016 May;195(5):1471-1473. doi: 10.1016/j.juro.2016.02.022. Epub 2016 Feb 10. No abstract available. PMID 27186728
- [Background] D'Amico AV, Chen MH, Renshaw A, Loffredo M, Kantoff PW. Long-term Follow-up of a Randomized Trial of Radiation With or Without Androgen Deprivation Therapy for Localized Prostate Cancer. JAMA. 2015 Sep 22-29;314(12):1291-3. doi: 10.1001/jama.2015.8577. No abstract available. PMID 26393854
- [Result] D'Amico AV, Manola J, Loffredo M, Renshaw AA, DellaCroce A, Kantoff PW. 6-month androgen suppression plus radiation therapy vs radiation therapy alone for patients with clinically localized prostate cancer: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):821-7. doi: 10.1001/jama.292.7.821. PMID 15315996
- [Result] Nguyen PL, Chen MH, Beard CJ, Suh WW, Choueiri TK, Efstathiou JA, Hoffman KE, Loffredo M, Kantoff PW, D'Amico AV. Comorbidity, body mass index, and age and the risk of nonprostate-cancer-specific mortality after a postradiation prostate-specific antigen recurrence. Cancer. 2010 Feb 1;116(3):610-5. doi: 10.1002/cncr.24818. PMID 19957321
- [Result] Nguyen PL, Chen MH, Beard CJ, Suh WW, Renshaw AA, Loffredo M, McMahon E, Kantoff PW, D'Amico AV. Radiation with or without 6 months of androgen suppression therapy in intermediate- and high-risk clinically localized prostate cancer: a postrandomization analysis by risk group. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):1046-52. doi: 10.1016/j.ijrobp.2009.06.038. Epub 2009 Oct 26. PMID 19864082
- [Result] Wo JY, Chen MH, Nguyen PL, Renshaw AA, Loffredo MJ, Kantoff PW, D'Amico AV. Evaluating the combined effect of comorbidity and prostate-specific antigen kinetics on the risk of death in men after prostate-specific antigen recurrence. J Clin Oncol. 2009 Dec 10;27(35):6000-5. doi: 10.1200/JCO.2009.23.6067. Epub 2009 Oct 26. PMID 19858385
- [Result] Nguyen PL, Chen MH, Renshaw AA, Loffredo M, Kantoff PW, D'Amico AV. Survival following radiation and androgen suppression therapy for prostate cancer in healthy older men: implications for screening recommendations. Int J Radiat Oncol Biol Phys. 2010 Feb 1;76(2):337-41. doi: 10.1016/j.ijrobp.2009.01.045. Epub 2009 Apr 22. PMID 19395186
- [Result] D'Amico AV, Chen MH, Renshaw AA, Loffredo M, Kantoff PW. Interval to testosterone recovery after hormonal therapy for prostate cancer and risk of death. Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):10-5. doi: 10.1016/j.ijrobp.2008.10.082. Epub 2009 Apr 22. PMID 19395184
- [Result] Tseng YD, Chen MH, Beard CJ, Martin NE, Orio PF, Loffredo M, Renshaw AA, Choueiri TK, Hu JC, Kantoff PW, D'Amico AV, Nguyen PL. Posttreatment prostate specific antigen nadir predicts prostate cancer specific and all cause mortality. J Urol. 2012 Jun;187(6):2068-73. doi: 10.1016/j.juro.2012.01.073. Epub 2012 Apr 11. PMID 22498212
- [Result] Chandra RA, Chen MH, Zhang D, Loffredo M, D'Amico AV. Evidence suggesting that obesity prevention measures may improve prostate cancer outcomes using data from a prospective randomized trial. Prostate Cancer. 2014;2014:478983. doi: 10.1155/2014/478983. Epub 2014 Feb 13. PMID 24693436
- [Result] Braunstein LZ, Chen MH, Loffredo M, Kantoff PW, D'Amico AV. Obesity and the Odds of Weight Gain following Androgen Deprivation Therapy for Prostate Cancer. Prostate Cancer. 2014;2014:230812. doi: 10.1155/2014/230812. Epub 2014 Apr 22. PMID 24864213
- [Derived] King MT, Chen MH, Collette L, Neven A, Bolla M, D'Amico AV. Association of Increased Prostate-Specific Antigen Levels After Treatment and Mortality in Men With Locally Advanced vs Localized Prostate Cancer: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2021 May 3;4(5):e2111092. doi: 10.1001/jamanetworkopen.2021.11092. PMID 33999161
- [Derived] Royce TJ, Chen MH, Wu J, Loffredo M, Renshaw AA, Kantoff PW, D'Amico AV. Surrogate End Points for All-Cause Mortality in Men With Localized Unfavorable-Risk Prostate Cancer Treated With Radiation Therapy vs Radiation Therapy Plus Androgen Deprivation Therapy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2017 May 1;3(5):652-658. doi: 10.1001/jamaoncol.2016.5983. PMID 28097317
- [Derived] Giacalone NJ, Wu J, Chen MH, Renshaw A, Loffredo M, Kantoff PW, D'Amico AV. Prostate-Specific Antigen Failure and Risk of Death Within Comorbidity Subgroups Among Men With Unfavorable-Risk Prostate Cancer Treated in a Randomized Trial. J Clin Oncol. 2016 Nov 1;34(31):3781-3786. doi: 10.1200/JCO.2016.68.4530. PMID 27601545
- [Derived] Kim MB, Chen MH, de Castro M, Loffredo M, Kantoff PW, D'Amico AV. Defining the optimal approach to the patient with postradiation prostate-specific antigen recurrence using outcome data from a prospective randomized trial. Cancer. 2013 Sep 15;119(18):3280-6. doi: 10.1002/cncr.28202. Epub 2013 Jun 24. PMID 23798006
- [Derived] D'Amico AV, Chen MH, Renshaw AA, Loffredo M, Kantoff PW. Androgen suppression and radiation vs radiation alone for prostate cancer: a randomized trial. JAMA. 2008 Jan 23;299(3):289-95. doi: 10.1001/jama.299.3.289. PMID 18212313